CLINICAL TRIAL: NCT02144610
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of AMG0001 in Subjects With Critical Limb Ischemia
Brief Title: Efficacy and Safety of AMG0001 in Subjects With Critical Limb Ischemia
Acronym: AGILITY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: AnGes USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG-CLI-0206; 2014-001129-34 (EudraCT Number)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Critical Limb Ischemia
Keywords: CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gene Therapy HGF Plasmid (AMG0001) (Experimental): Randomized subjects will receive 4 sets of intramuscular (IM) injections of HGF plasmid two weeks apart starting at Day 0 and again at Month 3 (first cycle) and at Month 9 and again at Month 12 (second cycle) in muscles of the affected lower limb.
  Interventions: Biological: HGF Plasmid (AMG0001)
- Placebo (Placebo Comparator): Randomized subjects will receive 4 sets of intramuscular (IM) injections of matching placebo two weeks apart starting at Day 0 and again at Month 3 (first cycle) and at Month 9 and again at Month 12 (second cycle) in muscles of the affected lower limb.
  Interventions: Biological: Matching Placebo

INTERVENTIONS:
Biological: HGF Plasmid (AMG0001) — IM
  Other Names: Beperminogene perplasmid (INN)
  Arms: Gene Therapy HGF Plasmid (AMG0001)
Biological: Matching Placebo — IM
  Arms: Placebo

SUMMARY:
Study to Evaluate the Efficacy and Safety of AMG0001 in Subjects with Critical Limb Ischemia.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, phase 3, multinational, multicenter study of AMG0001 (HGF plasmid) in subjects with Critical Limb Ischemia (CLI).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with CLI (Severe Rutherford 4 and Rutherford 5) who have:

   * No option for revascularization by endovascular intervention or surgical bypass

   or
   * Poor option (high risk) for revascularization by surgery and no option for an endovascular intervention (see Section 3.1 Study Population for full definition for appropriate inclusions).
2. Subjects 40-90 years of either gender who have signed an informed consent form either directly or through a legally authorized representative.
3. Subjects currently are taking a statin and an anti-platelet agent (e.g., clopidogrel, ticlopidine, aspirin, etc.) for 2 weeks or more prior to Day 0 as part of their standard of care, unless contraindicated. Subjects for whom these agents are contraindicated will have the reason for contraindication recorded in their case report form (CRF).
4. If female, the subjects must not be of child bearing potential, e.g., post-menopausal or surgically sterile.
5. If a male subject is of reproductive potential, he must agree to use an accepted and effective (barrier) form of birth control starting with the first dose of study product and continue for 12 weeks from the last dose of study product. This applies to both courses of treatment.
6. Subjects with a previous medical history of myocardial infarction and/or stroke should have adequate management of risk factors to prevent secondary occurrence. (See Section 4.2 Medical History for guidelines on appropriate secondary prevention.)
7. Subjects should have the ability to understand the requirements of the protocol and agree to return for the required study visits, assessments and follow up.

   * The index leg will be the leg with the greater severity of CLI disease. Entry requirements apply to the index leg. The index leg may also be referred to as the treated leg or affected leg in the text of this protocol or other study documents. If the subject has two legs that have the same Rutherford classification (severe Rutherford 4 or Rutherford 5) and are both eligible for treatment, the leg with greater disease severity (based on more extensive necrosis or more extensive/deeper ulceration(s), difference in ABI (ankle brachial index) or TBI (toe brachial index) ≥ 0.1, and/or more extensive vascular disease based on the angiogram) will be chosen as the index leg. If there is no clinical, hemodynamic or angiographic or other evidence to determine which leg has greater disease severity, the subject will be excluded from the study.
   * These entry criteria will be enforced (prior to randomization) by the Sponsor, as well as an Entry Committee who will review all relevant clinical data including but not limited to medical illness, CLI status, the findings of an angiogram, ulcer photographs and measurements and hemodynamic data.

Exclusion Criteria:

1. Subjects whose CLI status is unstable (spontaneous marked improvement or marked worsening during the screening period) or who have excessive tissue necrosis that is unlikely to benefit from medication, or those poor option subjects requiring immediate revascularization by surgery. Stability of the CLI status will be confirmed by the Principal Investigator prior to randomization and retrospectively reviewed by the Adjudication Committee.
2. Subjects who may require a major amputation (amputation at or above the ankle) within 4 weeks of Day 0 (± 4 weeks of Day 0).
3. Subjects with ulcers with exposure of tendons, osteomyelitis or uncontrolled infection or with the largest ulcer that is greater than 20 cm2 in area (>10 cm2 area if on the heel).
4. Subjects with purely neuropathic, or with venous ulcers.
5. Subjects in Rutherford 6 class.
6. Subjects who have had revascularization by surgery or angioplasty within 3 months, unless the procedure has failed based on the anatomy or the hemodynamic measurements.
7. Subjects with a diagnosis of Buerger's disease (Thrombo-angiitis Obliterans).
8. Subjects currently receiving immunosuppressive, chemo or radiation therapy.
9. Evidence or history of malignant neoplasm (clinical, laboratory or imaging) except for successfully excised basal cell or squamous cell carcinoma, or successfully excised early melanoma of the skin. Subjects, who had successful tumor resection or radio-chemotherapy of breast cancer more than 10 years prior to inclusion in the study, and with no recurrence, may be enrolled in the study. Subjects, who had successful tumor resection or radio-chemotherapy of all other tumor types and have been in remission for more than 5 years prior to inclusion in the study, and with no recurrence, may be enrolled in the study. A dermatological exam will have ruled out any skin cancer.
10. Subjects who have proliferative retinopathy, or moderate or severe non-proliferative retinopathy, from any cause (ETDRS Score > 35), clinically significant macular oedema or previous panretinal photocoagulation therapy (Results from the Early Treatment Diabetic Retinopathy Study. Ophthalmology May 1991 Supplement 98: 823-833).
11. Females of child-bearing potential defined as subjects that are not surgically sterile or post-menopausal.
12. Subjects with severe renal disease defined as significant renal dysfunction evidenced by an estimated creatinine clearance of <30 mL/minute (calculated using the Cockcroft Gault formula), or receiving chronic hemodialysis therapy.
13. Any co-morbid condition likely to interfere with assessment of safety or efficacy endpoints, acute cardiovascular events (i.e., CVA (cardiovascular accident), MI (myocardial infarction), etc.) within 3 months of treatment, or any disease that in the opinion of the Investigator may result in subject mortality in less than 3 months.
14. Subjects with known liver disease (e.g., hepatitis B or C or cirrhosis of the liver).
15. A subject with HIV, AIDS, severe uncontrolled inflammatory disease or severe uncontrolled autoimmune disease (e.g., ulcerative colitis, Crohn's disease, etc).
16. Subjects who have a significant psychiatric disorder or mental disability that could interfere with the subject's ability to provide informed consent or comply with study procedures.
17. Subjects with a current, uncorrected history of alcohol or substance abuse.
18. Diabetic subjects with an uncorrected HbA1c > 9.0% during the screening period.
19. Subjects that have been administered rhPDGF (e.g, becaplermin) or other growth factors locally within one month of randomization.
20. Subjects who have received another investigational drug within 30 days of randomization or have previously received any gene transfer therapy within 3 years of entering the study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Powell, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (59):
- United States (28):
  - Carondelet Heart and Vascular Institute, Tucson, Arizona
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - University of California, San Diego (UCSD), La Jolla, California
  - Alliance Research Centers, Laguna Hills, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Sarasota Memorial Hospital Clinical Research Center, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Harbin Clinic, LLC, Rome, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Peninsula Region Medical Center, Salisbury, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Luke's Hospital, Kansas City, Missouri
  - Kansas City Vascular P.C., Kansas City, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Oklahoma - Physicians Surgical Specialists, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - The Methodist Hospital Research Institute, Houston, Texas
- Belgium (3):
  - Antwerpen University Hospital, Edegem
  - Ziekenhuis Oost Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
- Jewish General Hospital, Montreal, Quebec, Canada
- Regionshospitalet Viborg, Viborg, Denmark
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- France (4):
  - Hopital Cardiologique - CHU Lille, Lille, Nord
  - CHU Amiens - Groupe Hospitalier Hopital Sud, Amiens
  - Hôpital Saint André, Bordeaux
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
- Hungary (11):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Belgyogyaszati Klinika, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bekes Megyei Pandy Kalman Korhaz Ersebeszet, Gyula
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz Altalanos- Mellkas es Ersebeszeti Osztaly, Kaposvár
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem AOK, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinika Központ, Szeged
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Universita Cattolica Policlinico Gemelli, Roma, Italy
- Netherlands (3):
  - Leiden Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (3):
  - Szpital Uniwersytecki nr 1 im. Dr A. Jurasza w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
- Karlkirurgiska Kliniken, Karolinska Universitetssjukhuset, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with critical limb ischemia from 69 sites across the United States, Canada, and Europe. The last patient completed in November 28, 2016.
Pre-assignment Details: Of the 98 subjects screened, 46 met the entry criteria and were randomized (1:1) into the study to receive AMG0001 or placebo as 4 sets of injections 2 weeks apart at Day 0, Month 3, Month 9, and Month 12.
Groups:
- Gene Therapy HGF Plasmid (AMG0001): Randomized subjects will receive 4 sets of intramuscular (IM) injections of hepatocyte growth factor (HGF) plasmid two weeks apart starting at Day 0 and again at Month 3 (first cycle) and at Month 9 and again at Month 12 (second cycle) in muscles of the affected lower limb, for a total of 16 sets of IM injections.
  Each set will be 8 IM injections; each IM injection contains 3 mL AMG0001.
  HGF Plasmid (AMG0001): IM
- Placebo: Randomized subjects will receive 4 sets of intramuscular (IM) injections of matching placebo two weeks apart starting at Day 0 and again at Month 3 (first cycle) and at Month 9 and again at Month 12 (second cycle) in muscles of the affected lower limb, for a total of 16 sets of IM injections.
  Each set will be 8 IM injections; each IM injection contains 3 mL placebo.
  Matching Placebo: IM
Period: Overall Study
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Started | 23 | 23
Completed | 0 | 1
Not Completed | 23 | 22
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Death | 2 | 2
Not completed — Study Discontinuation by Sponsor | 19 | 14
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Gene Therapy HGF Plasmid (AMG0001): Randomized subjects will receive 4 sets of intramuscular injections of HGF plasmid two weeks apart starting at Day 0 and again at Month 3 (first cycle) and at Month 9 and again at Month 12 (second cycle) in muscles of the affected lower limb.
  HGF Plasmid (AMG0001): IM
- Placebo: Randomized subjects will receive 4 sets of intramuscular injections of matching placebo two weeks apart starting at Day 0 and again at Month 3 (first cycle) and at Month 9 and again at Month 12 (second cycle) in muscles of the affected lower limb.
  Matching Placebo: IM
- Total: Total of all reporting groups
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (12) | 67 (9.79) | 67.3 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 17 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 18 | 21 | 39
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 2
  Belgium | 1 | 1 | 2
  Hungary | 8 | 6 | 14
  United States | 12 | 12 | 24
  Poland | 0 | 1 | 1
  France | 1 | 2 | 3
Past Tobacco Use [Count of Participants; unit: Participants]
  Yes | 14 | 18 | 32
  No | 9 | 5 | 14
Current Tobacco Use [Count of Participants; unit: Participants]
  Yes | 6 | 6 | 12
  No | 17 | 17 | 34
Alcohol Use [Count of Participants; unit: Participants]
  Yes | 8 | 6 | 14
  No | 15 | 17 | 32
Ulcer Present [Count of Participants; unit: Participants] | 11 | 13 | 24
Ischemic Rest Pain (cm) [Mean (Standard Deviation); unit: cm] — The severity of rest pain (based on the average over previous 7 days) recorded using the 10 cm visual analog scale (VAS).
  VAS is a 10-cm line (with score ranges 0 to 10), oriented horizontally; the left end of the line (0 mark) indicates "no pain"; the right end indicates "pain as bad as it can be."
  1. The subject is asked to mark a place on the line corresponding to the average pain intensity experienced in the last 7 days.
  2. The distance along the scale is converted into a numeric reading by measuring the distance of the subjects mark in cm from the beginning of the scale (the 0 mark). Population: Number analyzed in row differs from overall due to missing measurements.
  cm
    number analyzed (Participants) | 23 | 21 | 44
    (all) | 5.03 (2.92) | 6.04 (2.82) | 5.52 (2.89)
Ankle-brachial index (ABI) at baseline [Mean (Standard Deviation); unit: ratio] — The hemodynamic status of the affected lower limb was evaluated to confirm the critical limb ischemia (CLI) diagnosis and the subject's suitability for inclusion into the study.
  ABI < 0.8 indicates ischemia, ABI > 1.3 indicates incompressible vessel, normal range of ABI is >/= 0.8 and </=1.3. Population: Number analyzed in row differs from overall due to missing measurements.
  ratio
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 0.449 (0.1944) | 0.360 (0.2239) | 0.392 (0.218)
Toe-brachial index (TBI) at baseline [Mean (Standard Deviation); unit: ratio] — The hemodynamic status of the affected lower limb was evaluated to confirm the CLI diagnosis, and the subject's suitability for inclusion into the study. Population: Number analyzed in row differs from overall due to missing measurements.
  ratio
    number analyzed (Participants) | 21 | 18 | 39
    (all) | 0.134 (0.1280) | 0.167 (0.1660) | 0.149 (0.146)

OUTCOME MEASURES:

1. Primary Outcome: Major Amputation or Revascularization (of the Index Leg), All-cause Death, and Incidence of Stroke and Myocardial Infarction (MI)
Description: A frequency table for Day 0 to 6 months, Day 0 to 12 months and Day 0 to 18 months intervals by treatment group; the Fisher's Exact test was used for treatment comparison.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  0-6 Months (MI) | 1 | 0
  0-12 Months (MI) | 2 | 0
  0-18 Months (MI) | 2 | 0
  0-6 Months (Stroke) | 0 | 1
  0-12 Months (Stroke) | 1 | 1
  0-18 Months (Stroke) | 1 | 1
  0-6 Months (Major Amputation) | 5 | 7
  0-12 Months (Major Amputation) | 6 | 7
  0-18 Months (Major Amputation) | 6 | 7
  0-6 Months (Revascularization) | 3 | 2
  0-12 Months (Revascularization) | 6 | 3
  0-18 Months (Revascularization) | 6 | 3
  0-6 Months (All-cause Death) | 0 | 1
  0-12 Months (All-cause Death) | 2 | 2
  0-18 Months (All-cause Death) | 3 | 2
  0-6 Months (Major Amputation or Death) | 5 | 8
  0-12 Months (Major Amputation or Death) | 7 | 9
  0-18 Months (Major Amputation or Death) | 8 | 9
  0-6 Months (Major Amputation or Revascularization) | 7 | 9
  0-12 Month (Major Amputation or Revascularization) | 11 | 10
  0-18 Month (Major Amputation or Revascularization) | 11 | 10
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; MI at 0-6 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; MI at 0-12 Months; Test type: Superiority or Other; p = 0.4889, Fisher Exact
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; MI at 0-18 Months; Test type: Superiority or Other; p = 0.4889, Fisher Exact
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Stroke at 0-6 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Stroke at 0-12 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Stroke at 0-18 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 7: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Major amputation at 0-6 Months; Test type: Superiority or Other; p = 0.7381, Fisher Exact
Statistical Analysis 8: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Major amputation at 0-12 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 9: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Major amputation at 0-18 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 10: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Revascularization at 0-6 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 11: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Revascularization at 0-12 Months; Test type: Superiority or Other; p = 0.4591, Fisher Exact
Statistical Analysis 12: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Revascularization at 0-18 Months; Test type: Superiority or Other; p = 0.4591, Fisher Exact
Statistical Analysis 13: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; All-cause death at 0-6 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 14: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; All-cause death at 0-12 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 15: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; All-cause death at 0-18 Months; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 16: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; 0-6 Months (Major Amputation or Death); Test type: Superiority or Other; p = 0.5136, Fisher Exact
Statistical Analysis 17: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; 0-12 Months (Major Amputation or Death); Test type: Superiority or Other; p = 0.7575, Fisher Exact
Statistical Analysis 18: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; 0-18 Months (Major Amputation or Death); Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 19: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; 0-6 Months (Major Amputation or Revascularization); Test type: Superiority or Other; p = 0.7575, Fisher Exact
Statistical Analysis 20: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; 0-12 Months (Major Amputation or Revascularization); Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 21: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; 0-18 Months (Major Amputation or Revascularization); Test type: Superiority or Other; p > 0.999, Fisher Exact

2. Primary Outcome: Change in Ischemic Rest Pain (in the Index Leg) From Baseline Using a 10 cm Visual Analog Scale (VAS) Scale
Description: The severity of rest pain (based on the average over previous 7 days) recorded using the 10 cm visual analog scale (VAS).
  VAS is a 10-cm line (with score ranges 0 to 10), oriented horizontally; the left end of the line (0 mark) indicates "no pain"; the right end indicates "pain as bad as it can be."
  1. The subject is asked to mark a place on the line corresponding to the average pain intensity experienced in the last 7 days.
  2. The distance along the scale is converted into a numeric reading by measuring the distance of the subjects mark in cm from the beginning of the scale (the 0 mark).
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 19 | 16
score on a scale
  Change from Baseline at Month 3: number analyzed (Participants) | 18 | 16
  Change from Baseline at Month 3 | 0.40 (2.310) | -0.79 (2.889)
  Change from Baseline at Month 6: number analyzed (Participants) | 14 | 10
  Change from Baseline at Month 6 | 0.20 (3.002) | -1.65 (2.704)
  Change from Baseline at Month 9: number analyzed (Participants) | 11 | 5
  Change from Baseline at Month 9 | -0.15 (2.281) | -0.90 (2.801)
  Change from Baseline at Month 12: number analyzed (Participants) | 8 | 3
  Change from Baseline at Month 12 | -2.39 (2.156) | 0.00 (0.200)
  Change from Baseline at Month 15: number analyzed (Participants) | 3 | 2
  Change from Baseline at Month 15 | -0.80 (1.825) | 2.40 (1.980)
  Change from Baseline at LOCF | -1.61 (2.863) | -0.20 (3.087)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 3; Test type: Superiority or Other; p = 0.514, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 6; Test type: Superiority or Other; p = 0.445, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 9; Test type: Superiority or Other; p = 0.863, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 12; Test type: Superiority or Other; p = 0.111, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 15; Test type: Superiority or Other; p = 0.153, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at last observation carried forward (LOCF); Test type: Superiority or Other; p = 0.002, ANCOVA

3. Primary Outcome: Ulcer Improvement
Description: A table showing the number of subjects with complete healing of the target ulcer by treatment. Ulcer healing of the largest ulcer on the index limb was assessed clinically by the Principal Investigator by direct visual inspection at each study visit. If the largest ulcer on the index leg was considered completely healed, photographs of the healed ulcer area was captured. If an ulcer healed completely during the study period, the ulcer was re-evaluated 2 weeks later to confirm it has remained healed. Confirmation of complete ulcer healing was made by an outside physician unconnected with the study and nominated for this purpose.
Time Frame: 18 months
Population: The number of participants analyzed are those that have an ulcer on the index leg at the time of enrollment (n=11 in HGF plasmid group, n=13 in placebo group).
Measure: Count of Participants; unit: Participants
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 11 | 13
Participants
  Baseline and up to Month 6 | 2 | 1
  Baseline and up to Month 12 | 3 | 1
  Baseline and up to Month 18 | 3 | 1

4. Primary Outcome: VAS Improvement
Description: A table showing the number of subjects with improvement in VAS (≥ 20 mm) by treatment.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  Baseline and up to Month 6 | 4 | 6
  Baseline and up to Month 12 | 9 | 6
  Baseline and up to Month 18 | 9 | 6

5. Primary Outcome: Hemodynamic Measurements - Mean Change From Baseline in Brachial (Right/Left) Systolic Pressure
Description: Summary statistics were provided for baseline and change from baseline for right/left brachial systolic pressure by visit and treatment (only subjects with non-missing baseline and visit values). A two-way analysis of covariance (ANCOVA) with treatment and region as fixed factors and baseline as a covariate were performed for each visit and LOCF.
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 19 | 15
mmHg
  Change from Baseline at Month 3 (right): number analyzed (Participants) | 18 | 15
  Change from Baseline at Month 3 (right) | 0.7 (27.27) | 2.4 (18.78)
  Change from Baseline at Month 6 (right): number analyzed (Participants) | 14 | 9
  Change from Baseline at Month 6 (right) | -2.4 (23.49) | 0.7 (33.58)
  Change from Baseline at Month 9 (right): number analyzed (Participants) | 9 | 5
  Change from Baseline at Month 9 (right) | 2.3 (14.50) | -7.2 (26.52)
  Change from Baseline at Month 12 (right): number analyzed (Participants) | 8 | 4
  Change from Baseline at Month 12 (right) | -5.8 (16.76) | 5.0 (15.60)
  Change from Baseline at Month 15 (right): number analyzed (Participants) | 3 | 3
  Change from Baseline at Month 15 (right) | 5.7 (22.81) | 13.0 (6.08)
  Change from Baseline at Month 18 (right): number analyzed (Participants) | 0 | 1
  Change from Baseline at Month 18 (right) |  | 23.0
  Change from Baseline at LOCF (right) | -2.3 (24.36) | 8.2 (23.94)
  Change from Baseline at Month 3 (left): number analyzed (Participants) | 16 | 14
  Change from Baseline at Month 3 (left) | 7.9 (27.37) | -5.7 (22.24)
  Change from Baseline at Month 6 (left): number analyzed (Participants) | 14 | 9
  Change from Baseline at Month 6 (left) | -1.1 (28.61) | -15.8 (30.04)
  Change from Baseline at Month 9 (left): number analyzed (Participants) | 9 | 5
  Change from Baseline at Month 9 (left) | -0.8 (14.52) | -25.8 (30.78)
  Change from Baseline at Month 12 (left): number analyzed (Participants) | 8 | 3
  Change from Baseline at Month 12 (left) | 0.6 (14.00) | 10.0 (11.36)
  Change from Baseline at Month 15 (left: number analyzed (Participants) | 3 | 2
  Change from Baseline at Month 15 (left | 4.7 (21.01) | -18.5 (38.89)
  Change from Baseline at Month 18 (left): number analyzed (Participants) | 0 | 1
  Change from Baseline at Month 18 (left) |  | -2.0
  Change from Baseline at LOCF (left) | 2.6 (26.68) | -0.9 (19.20)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 3 (right brachial); Test type: Superiority or Other; p = 0.733, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 6 (right brachial); Test type: Superiority or Other; p = 0.808, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 9 (right brachial); Test type: Superiority or Other; p = 0.487, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 12 (right brachial); Test type: Superiority or Other; p = 0.216, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 15 (right brachial); Test type: Superiority or Other; p = 0.896, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at last observation carried forward (LOCF) (right brachial); Test type: Superiority or Other; p = 0.167, ANCOVA
Statistical Analysis 7: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 3 (left brachial); Test type: Superiority or Other; p = 0.378, ANCOVA
Statistical Analysis 8: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 6 (left brachial); Test type: Superiority or Other; p = 0.390, ANCOVA
Statistical Analysis 9: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 9 (left brachial); Test type: Superiority or Other; p = 0.521, ANCOVA
Statistical Analysis 10: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 12 (left brachial); Test type: Superiority or Other; p = 0.044, ANCOVA
Statistical Analysis 11: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at Month 15 (left brachial); Test type: Superiority or Other; p = 0.423, ANCOVA
Statistical Analysis 12: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from baseline at LOCF (left brachial); Test type: Superiority or Other; p = 0.989, ANCOVA

6. Primary Outcome: Hemodynamic Measurements - Mean Change From Baseline in Ankle (Dorsalis Pedis/Posterior Tibial) Systolic Pressure
Description: Summary statistics were provided for baseline and change from baseline for ankle systolic pressure measured at dorsalis pedis and posterior tibial by visit and treatment (only subjects with non-missing baseline and visit values). A two-way analysis of covariance (ANCOVA) with treatment and region as fixed factors and baseline as a covariate were performed for each visit and LOCF.
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 14 | 12
mmHg
  Change from Baseline at Month 3 (Dorsalis Pedis): number analyzed (Participants) | 12 | 12
  Change from Baseline at Month 3 (Dorsalis Pedis) | 4.2 (35.66) | 11.2 (30.15)
  Change from Baseline at Month 6 (Dorsalis Pedis): number analyzed (Participants) | 10 | 8
  Change from Baseline at Month 6 (Dorsalis Pedis) | 12.7 (19.96) | 9.9 (22.73)
  Change from Baseline at Month 9 (Dorsalis Pedis): number analyzed (Participants) | 5 | 5
  Change from Baseline at Month 9 (Dorsalis Pedis) | 3.4 (40.59) | 3.0 (57.86)
  Change from Baseline at Month 12 (Dorsalis Pedis): number analyzed (Participants) | 5 | 3
  Change from Baseline at Month 12 (Dorsalis Pedis) | 59.4 (47.00) | 12.0 (15.62)
  Change from Baseline at Month 15 (Dorsalis Pedis): number analyzed (Participants) | 2 | 1
  Change from Baseline at Month 15 (Dorsalis Pedis) | 18.5 (10.61) | 3.0
  Change from Baseline at LOCF (Dorsalis Pedis) | 32.9 (41.55) | 16.7 (34.25)
  Change from Baseline at Month 3 (Posterior Tibial): number analyzed (Participants) | 13 | 10
  Change from Baseline at Month 3 (Posterior Tibial) | 15.2 (35.02) | 16.1 (31.81)
  Change from Baseline at Month 6 (Posterior Tibial): number analyzed (Participants) | 8 | 6
  Change from Baseline at Month 6 (Posterior Tibial) | 28.4 (28.32) | 19.2 (37.04)
  Change from Baseline at Month 9 (Posterior Tibial): number analyzed (Participants) | 4 | 4
  Change from Baseline at Month 9 (Posterior Tibial) | 4.5 (24.64) | -3.5 (15.50)
  Change from Baseline atMonth 12 (Posterior Tibial): number analyzed (Participants) | 4 | 3
  Change from Baseline atMonth 12 (Posterior Tibial) | 45.0 (28.86) | 4.3 (5.86)
  Change from Baseline atMonth 15 (Posterior Tibial): number analyzed (Participants) | 2 | 1
  Change from Baseline atMonth 15 (Posterior Tibial) | 40.5 (51.62) | -10.0
  Change from Baseline at LOCF (Posterior Tibial): number analyzed (Participants) | 12 | 11
  Change from Baseline at LOCF (Posterior Tibial) | 35.1 (33.97) | 13.2 (24.98)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 3 (Dorsalis Pedis); Test type: Superiority or Other; p = 0.803, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 6 (Dorsalis Pedis); Test type: Superiority or Other; p = 0.668, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 9 (Dorsalis Pedis); Test type: Superiority or Other; p = 0.789, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 12 (Dorsalis Pedis); Test type: Superiority or Other; p = 0.280, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at LOCF (Dorsalis Pedis); Test type: Superiority or Other; p = 0.324, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 3 (Posterior Tibial); Test type: Superiority or Other; p = 0.759, ANCOVA
Statistical Analysis 7: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 6 (Posterior Tibial); Test type: Superiority or Other; p = 0.414, ANCOVA
Statistical Analysis 8: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 9 (Posterior Tibial); Test type: Superiority or Other; p = 0.886, ANCOVA
Statistical Analysis 9: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 12 (Posterior Tibial); Test type: Superiority or Other; p = 0.114, ANCOVA
Statistical Analysis 10: Comparison: Gene Therapy HGF Plasmid (AMG0001); Change from Baseline at LOCF (Posterior Tibial); Test type: Superiority or Other; p = 0.051, ANCOVA

7. Primary Outcome: Hemodynamic Measurements - Mean Change From Baseline in Toe Systolic Pressure
Description: Summary statistics were provided for baseline and change from baseline for toe systolic pressure by visit and treatment (only subjects with non-missing baseline and visit values). A two-way analysis of covariance (ANCOVA) with treatment and region as fixed factors and baseline as a covariate were performed for each visit and LOCF.
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 16 | 11
mmHg
  Change from Baseline at Month 3: number analyzed (Participants) | 15 | 10
  Change from Baseline at Month 3 | 4.4 (19.96) | -9.9 (25.07)
  Change from Baseline at Month 6: number analyzed (Participants) | 11 | 8
  Change from Baseline at Month 6 | 19.5 (18.44) | -6.3 (33.76)
  Change from Baseline at Month 9: number analyzed (Participants) | 9 | 4
  Change from Baseline at Month 9 | 20.7 (20.38) | 29.3 (28.79)
  Change from Baseline at Month 12: number analyzed (Participants) | 6 | 3
  Change from Baseline at Month 12 | 34.8 (37.38) | 39.3 (19.63)
  Change from Baseline at Month 15: number analyzed (Participants) | 3 | 2
  Change from Baseline at Month 15 | 16.0 (33.05) | 6.5 (9.19)
  Change from Baseline at Month 18: number analyzed (Participants) | 0 | 1
  Change from Baseline at Month 18 |  | 14.0
  Change from Baseline at LOCF | 18.5 (32.51) | -2.9 (30.04)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 3; Test type: Superiority or Other; p = 0.211, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 6; Test type: Superiority or Other; p = 0.036, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 9; Test type: Superiority or Other; p = 0.725, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 12; Test type: Superiority or Other; p = 0.468, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 15; Test type: Superiority or Other; p = 0.854, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at LOCF; Test type: Superiority or Other; p = 0.233, ANCOVA

8. Primary Outcome: Hemodynamic Measurements - Mean Change From Baseline in ABI of Index Leg
Description: Summary statistics were provided for baseline and change from baseline for calculated ABI by visit and treatment (only subjects with non-missing baseline and visit values). A two-way analysis of covariance (ANCOVA) with treatment and region as fixed factors and baseline as a covariate were performed for each visit and LOCF.
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 16 | 15
ratio
  Change from Baseline at Month 3: number analyzed (Participants) | 14 | 14
  Change from Baseline at Month 3 | -0.009 (0.2612) | 0.105 (0.1661)
  Change from Baseline at Month 6: number analyzed (Participants) | 11 | 10
  Change from Baseline at Month 6 | 0.097 (0.0920) | 0.028 (0.2257)
  Change from Baseline at Month 9: number analyzed (Participants) | 6 | 5
  Change from Baseline at Month 9 | 0.098 (0.1001) | 0.246 (0.3272)
  Change from Baseline at Month 12: number analyzed (Participants) | 6 | 4
  Change from Baseline at Month 12 | 0.303 (0.3481) | 0.098 (0.0964)
  Change from Baseline at Month 15: number analyzed (Participants) | 3 | 2
  Change from Baseline at Month 15 | -0.077 (0.2101) | 0.090 (0.1556)
  Change from Baseline at LOCF | 0.115 (0.3662) | 0.111 (0.1855)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 3; Test type: Superiority or Other; p = 0.268, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 6; Test type: Superiority or Other; p = 0.320, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 9; Test type: Superiority or Other; p = 0.315, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 12; Test type: Superiority or Other; p = 0.327, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 15; Test type: Superiority or Other; p = 0.643, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at LOCF; Test type: Superiority or Other; p = 0.740, ANCOVA

9. Primary Outcome: Hemodynamic Measurements - Mean Change From Baseline in TBI of Index Leg
Description: Summary statistics were provided for baseline and change from baseline for calculated TBI by visit and treatment (only subjects with non-missing baseline and visit values). A two-way analysis of covariance (ANCOVA) with treatment and region as fixed factors and baseline as a covariate were performed for each visit and LOCF.
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 17 | 14
ratio
  Change from Baseline at Month 3: number analyzed (Participants) | 16 | 12
  Change from Baseline at Month 3 | 0.024 (0.1661) | -0.078 (0.1536)
  Change from Baseline at Month 6: number analyzed (Participants) | 12 | 9
  Change from Baseline at Month 6 | 0.133 (0.1398) | -0.037 (0.2175)
  Change from Baseline at Month 9: number analyzed (Participants) | 9 | 5
  Change from Baseline at Month 9 | 0.134 (0.1493) | 0.112 (0.1747)
  Change from Baseline at Month 12: number analyzed (Participants) | 7 | 4
  Change from Baseline at Month 12 | 0.303 (0.2945) | 0.238 (0.2045)
  Change from Baseline at Month 15: number analyzed (Participants) | 3 | 2
  Change from Baseline at Month 15 | 0.110 (0.2261) | 0.035 (0.0495)
  Change from Baseline at Month 18: number analyzed (Participants) | 0 | 1
  Change from Baseline at Month 18 |  | 0.070
  Change from Baseline at LOCF | 0.168 (0.2692) | -0.044 (0.1846)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 3; Test type: Superiority or Other; p = 0.147, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 6; Test type: Superiority or Other; p = 0.032, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 9; Test type: Superiority or Other; p = 0.709, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 12; Test type: Superiority or Other; p = 0.771, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 15; Test type: Superiority or Other; p = 0.830, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at LOCF; Test type: Superiority or Other; p = 0.033, ANCOVA

10. Primary Outcome: Changes in the Quality of Life Using the Vascular Quality of Life Questionnaire (VascuQol) Over 18 Months
Description: The VascuQol contains 5 domains (pain, symptom, activities, social, and emotional functioning); responses were scored from 0 (lowest QOL, death) to 7 (best QOL, maximum health).
  Responses were averaged for composite overall and domain-specific scores, giving equal weight to each question and domain. The composite overall is the average of domain-specific scores.
  Responses after revascularization or major amputation were included in the analysis. In the event of death, subjects were scored as 0. For the effect of treatment on individual domains, pain, symptoms, and activities were considered the most important of the 5 domains.
  Summary statistics were provided for baseline and change from baseline by visit and treatment for VascuQol, including subscore, for subjects who had a non-missing value at both baseline and the specific visit. A two-way ANCOVA with treatment and region as fixed factors and baseline as a covariate were performed for each visit and LOCF.
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale
  Pain (LOCF): number analyzed (Participants) | 19 | 18
  Pain (LOCF) | 1.46 (1.158) | 0.83 (1.557)
  Symptom (LOCF): number analyzed (Participants) | 19 | 18
  Symptom (LOCF) | 0.79 (1.475) | 0.71 (1.468)
  Activities (LOCF): number analyzed (Participants) | 19 | 18
  Activities (LOCF) | 0.59 (0.950) | 0.66 (0.981)
  Social (LOCF): number analyzed (Participants) | 19 | 18
  Social (LOCF) | 0.53 (1.086) | 0.39 (1.852)
  Emotional Functioning (LOCF) | 0.77 (1.247) | 0.83 (1.458)
  Composite Overall (LOCF) | 0.81 (0.843) | 0.74 (1.068)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Pain (LOCF); Test type: Superiority or Other; p = 0.105, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Symptom (LOCF); Test type: Superiority or Other; p = 0.557, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Activities (LOCF); Test type: Superiority or Other; p = 0.940, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Social (LOCF); Test type: Superiority or Other; p = 0.905, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Emotional Functioning (LOCF); Test type: Superiority or Other; p = 0.782, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Composite Overall (LOCF); Test type: Superiority or Other; p = 0.802, ANCOVA

11. Primary Outcome: Changes in the Quality of Life From Baseline Using the EQ-5D-5L Over 18 Months
Description: The EQ-5D-5L descriptive system covers 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5); death was coded as a worst case.
  The EQ-5D-5L health state for each subject, referred to as a 5 digit code that combines 1 level from each of the 5 dimensions, was converted into a single index value using a published weighing system. The index value ranges from -0.109 to 1, where 1 indicates no problems in all 5 dimensions, and is reduced when a patient reports increasing problems.
  Summary statistics were provided for baseline and change from baseline by visit and treatment for EQ-5D-5L, including subscore, for subjects who had a non-missing value at both baseline and the specific visit. A two-way ANCOVA with treatment and region as fixed factors and baseline as a covariate were performed for each visit and LOCF.
Time Frame: 18 months
Population: The number analyzed in one or more rows differs from overall number analyzed due to early discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 20 | 19
score on a scale
  Change from Baseline at Month 3: number analyzed (Participants) | 17 | 18
  Change from Baseline at Month 3 | 0.03 (0.130) | 0.03 (0.149)
  Change from Baseline at Month 6: number analyzed (Participants) | 14 | 13
  Change from Baseline at Month 6 | 0.01 (0.127) | 0.04 (0.114)
  Change from Baseline at Month 9: number analyzed (Participants) | 12 | 7
  Change from Baseline at Month 9 | -0.06 (0.168) | 0.07 (0.092)
  Change from Baseline at Month 12: number analyzed (Participants) | 8 | 5
  Change from Baseline at Month 12 | 0.08 (0.193) | 0.08 (0.097)
  Change from Baseline at Month 15: number analyzed (Participants) | 3 | 3
  Change from Baseline at Month 15 | -0.03 (0.043) | 0.05 (0.156)
  Change from Baseline at Month 18: number analyzed (Participants) | 0 | 1
  Change from Baseline at Month 18 |  | -0.02
  Change from Baseline at LOCF | 0.04 (0.194) | 0.03 (0.153)
Statistical Analysis 1: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 3; Test type: Superiority or Other; p = 0.941, ANCOVA
Statistical Analysis 2: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 6; Test type: Superiority or Other; p = 0.584, ANCOVA
Statistical Analysis 3: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 9; Test type: Superiority or Other; p = 0.100, ANCOVA
Statistical Analysis 4: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 12; Test type: Superiority or Other; p = 0.916, ANCOVA
Statistical Analysis 5: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at Month 15; Test type: Superiority or Other; p = 0.486, ANCOVA
Statistical Analysis 6: Comparison: Gene Therapy HGF Plasmid (AMG0001) vs Placebo; Change from Baseline at LOCF; Test type: Superiority or Other; p = 0.835, ANCOVA

12. Post Hoc Outcome: Time to Major Amputation (of the Index Leg) or All-cause Death
Description: The median time to major amputation or death was analyzed over the duration of the study as a post-hoc analysis; all reports of major amputation or death were included in this post hoc analysis, irrespective of pre-defined study windows.
Time Frame: Month 36
Population: Subjects who had a major amputation or died during the study
Measure: Median (Full Range); unit: Days
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
Number analyzed (Participants) | 8 | 10
Days | 505 [0 to 528] | 381 [0 to 539]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were documented from the start of the first dose of study product (Day 0) to the end of the follow-up period (Month 18).
Arm/Group | Gene Therapy HGF Plasmid (AMG0001) | Placebo
All-Cause Mortality (participants affected / at risk) | 3/23 | 2/23
Serious Adverse Events (participants affected / at risk) | 7/23 | 9/23
Other Adverse Events (participants affected / at risk) | 5/23 | 7/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gene Therapy HGF Plasmid (AMG0001) (N=23) | Placebo (N=23)
suicidal ideation (Psychiatric disorders) | 1 | 0
pneumonia (Infections and infestations) | 1 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
angina unstable (Cardiac disorders) | 1 | 0
acute myocardial infarction (Cardiac disorders) | 2 | 0
multiple organ dysfunction syndrome (General disorders) | 1 | 0
cerebrovascular accident (Nervous system disorders) | 1 | 1
hypotension (Vascular disorders) | 1 | 0
cardiac failure congestive (Cardiac disorders) | 1 | 1
non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
anaemia (Blood and lymphatic system disorders) | 1 | 0
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
cardiac arrest (Cardiac disorders) | 0 | 1
bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
device related infection (Infections and infestations) | 0 | 1
vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
fall (Injury, poisoning and procedural complications) | 0 | 1
laceration (Injury, poisoning and procedural complications) | 0 | 1
sepsis (Infections and infestations) | 0 | 1
hip fracture (Injury, poisoning and procedural complications) | 0 | 1
carotid artery occlusion (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gene Therapy HGF Plasmid (AMG0001) (N=23) | Placebo (N=23)
urinary tract infection (Infections and infestations) | 3 | 1
nasopharyngitis (Infections and infestations) | 2 | 1
nausea (Gastrointestinal disorders) | 0 | 3
constipation (Gastrointestinal disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Because of early termination of study due to low subject enrollment, subject exposure to study treatment and the duration were highly variable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No